CLINICAL TRIAL: NCT04625829
Title: Anthropological Survey on the Use of Essential Oils (EOs) by Cystic Fibrosis Patients: a Quantitative and Qualitative Approach
Acronym: AROMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.303; 2020-A02375-34 (Other: ID RCB)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Mucoviscidosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients and parents of patients will be asked to answer a questionnaire on paper or online, by the CRCMs and through communication campaigns distributed by the association Vaincre La Mucoviscidose (VLM).

This questionnaire includes about fifty items that will take 5 to 12 minutes to complete. The study aims to interview 250 patients / parents of patients, users and non-users of essential oils.

Thirty patients or volunteer parents will then meet with a health anthropologist for qualitative interviews to document very precisely the modalities of use of essential oils: which ones, at what dose, advised by whom, the dedicated budget. Relationships with CRCM doctors, the effects felt, the side effects will also be explored.

The global data of the two phases will be integrated and put into perspective with the scientific data currently available on essential oils.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patient or parent of a child with cystic fibrosis

Exclusion Criteria:

* patient who refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cystic fibrosis patient
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of use of the different EO by the patients who answered the questionnaire | through study completion, an average of 1 year
  Frequency of use of the different EO by the patients who answered the questionnaire

IPD SHARING:
Plan to Share IPD: No